CLINICAL TRIAL: NCT06068088
Title: Preliminary Survey of Dietary Practices and Nutritional Status of Patients Treated With Radiochemotherapy for Non-small Cell Lung Carcinoma
Brief Title: Dietary Practices and Locally Advanced Lung Cancer (LUNGDIET)
Acronym: LUNGDIET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230706; IDRCB 2023-A00329-36 (Other: Agence nationale de sécurité du médicament et des produits de santé); 23.01988.000202 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2023-08-30; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Radiochemotherapy; Fasting; Special diet
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fasting | interventions — Blood Specimen Collection; Nutrition Assessment; Referral and Consultation; Nutritionists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Participating patients from 5 radiotherapy center of AP-HP
  Interventions: Behavioral: Self-administered survey at hospital
- Cohort B: Participating patients from the european hospital Georges-Pompidou
  Interventions: Behavioral: Self-administered survey at hospital; Biological: Blood sample for nutritional assessment; Other: Consultation with nutritionist doctor and dietician

INTERVENTIONS:
Behavioral: Self-administered survey at hospital — Self-administered survey on the food practices of the patient Completion before the beginning of chemoradiotherapy
Biological: Blood sample for nutritional assessment — 15 ml of blood sampled during nutritional examination before the beginning and during the month following the end of chemoradiotherapy
  Groups: Cohort B
Other: Consultation with nutritionist doctor and dietician — Before the beginning and during the month following the end of chemoradiotherapy Consultation of approximatively one hour
  Groups: Cohort B

SUMMARY:
In recent years, fasting or the use of special diets (ketogenic, high protein, etc.), whether or not associated with food supplements, have increased substantially, particularly in oncology with the idea of improving for some of them, the tolerance of the proposed treatments, in particular emetogenic chemotherapy, or even to improve the prognosis. Although there are preclinical data on cell cultures and in rats, the clinical data supporting these practices are very fragmented, with few trials carried out and only including small cohorts, mainly in the context of breast cancers. It is therefore very difficult to respond objectively to patients asking the question of the merits of these changes in dietary practices in the management of their cancer.

The investigators want to carry out an inventory of the dietary practices of participating patients and their potential interest in fasting or special diets by means of a self-administered survey completed by the patient at diagnosis before treatment. This semi-quantitative self-administered survey (answers in never / sometimes / regularly / systematically) was developed by the nutrition and radiotherapy team of the Georges-Pompidou European Hospital because there was no validated medical questionnaire on fasting or the use of special diets in oncology

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented inoperable stage III non-small cell lung carcinoma (no metastasis)
* Treatment with curative intent including thoracic radiotherapy and at least one cycle of concomitant chemotherapy
* Patient informed and having signed the consent

Exclusion Criteria:

* Sequential radiochemotherapy
* Metastatic forms from the outset
* Ear, nose, and throat (ENT) or digestive pathologies interfering with normal oral nutrition
* Other concurrent or pre-existing cancer for less than 5 years at the diagnosis of bronchial cancer
* Patient under guardianship or curatorship
* Patient with cognitive impairment
* Patient not affiliated with a social security
* Patient under state medical help from french government
* Radiotherapy performed outside the AP-HP for cohort A and outside the HEGP for cohort B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is aimed at patients treated with radiochemotherapy for non-small cell lung cancer localized in thorax. The choice of this population is based on its frequency, its clinical homogeneity, the prospect of a curative treatment but with a clearly improvable prognosis and the absence of published data on the subject.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Inventory of the dietary practices | 1 to 15 days
  Inventory of the dietary practices of participating patients and their potential interest in fasting or special diets by means of a self-administered survey completed by the patient at diagnosis before treatment. Determination of the proportions of patients who have already followed or respond favorably to the idea of fasting and/or a particular diet. The survey is semi-quantitative.

SECONDARY OUTCOMES:
Evaluate the nutritional status of patients before treatement with radiochemotherapy for non-small cell lung cancer located in the thorax. | 3 month
  Descriptive analysis of the nutritional status of the population before the start of radiochemotherapy.
Evaluate the nutritional status of patients in the month following the radiochemotherapy for non-small cell lung cancer located in the thorax. | 3 month
  Descriptive analysis of the nutritional status of the population in the month following the end of radiochemotherapy.
Evaluate the evolution of nutritional status in the population of the study | 3 month
  Descriptive analysis of the evolution (deterioration, stability, improvement) of the nutritional status of the population before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of total cholesterol in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter total cholesterol (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of High Density Lipoprotein (HDL) in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter High Density Lipoprotein (HDL) (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of Low Density Lipoprotein (LDL) in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter Low Density Lipoprotein (LDL) (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of triglycerides in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter triglycerides (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of uricemia in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter uricemia (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of fasting glucose in the population. | 3 month
  Descriptive analysis of the evolution of the metabolic parameter fasting glucose (mmol/L) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of Glycated hemoglobin (HbA1C) in the population | 3 month
  Descriptive analysis of the evolution of the metabolic parameter Glycated hemoglobin (HbA1C) (%) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of the index homeostasis model assessment (HOMA) in the population | 3 month
  Descriptive analysis of the evolution of the index HOMA (no unit) before the start of radiochemotherapy and in the month following the end of it.
Evaluate the evolution of Vitamin D in the population | 3 month
  Descriptive analysis of the evolution of the metabolic parameter vitamin D (ng/L) before the start of radiochemotherapy and in the month following the end of it.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine DURDUX, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).